CLINICAL TRIAL: NCT03191006
Title: Therapeutic Effects of Physical Function and Balance of Customized Insoles on Children With Developmental Delays
Brief Title: Effects of Insoles on Children With Developmental Delays
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Principal Investigator, Ru-Lan Hsieh, Professor, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SKH-8302-106-DR-28.
Record Dates: First submitted 2017-06-11; First posted 2017-06-19 (Actual); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Developmental Delay
Keywords: effect; insoles; children
MeSH Terms: conditions — Learning Disabilities

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group: MEI BIN insoles (Active Comparator): Participants in the study group will be prescribed with a pair of customized insoles (MEI BIN) to keep the subtalar joint in neutral position, for 12 weeks.
  Interventions: Device: MEI BIN insoles
- control group: without MEI BIN insoles (No Intervention): Participants in this control group will not receive a pair of customized insoles (MEI BIN) to keep the subtalar joint in neutral position, for 12 weeks.

INTERVENTIONS:
Device: MEI BIN insoles — insoles
  Arms: study group: MEI BIN insoles

SUMMARY:
Using double blind, randomized controlled design to investigate the short-term therapeutic effects of function of customized insoles on children with developmental delays

DETAILED DESCRIPTION:
A total of 52 children with developmental delays will be enrolled. The participants will be randomized into two groups, including study group (with insoles) and control group (without insoles).

The participants in the study group will be evaluated at baseline, that is before the customized insoles are prescribed. All of evaluations, including physical function, balance, and quality of life will be re-evaluated up to 12 weeks after insoles wearing.

The control group will be evaluated at the baseline and up to 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* developmental delays

Exclusion Criteria:

* age less than 3 years old or older than 10 years old normal development

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Estimated)
Dates: Start 2017-06-24 (Estimated); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline functional performance (scores) at 12 weeks | baseline and up to 12 weeks
  Pediatric Outcome Data Collection Instrument

SECONDARY OUTCOMES:
change from baseline physical function (time) at 12 weeks | baseline and up to 12 weeks
  time of stair climbing, timed up and go, walking on level ground
change from baseline balance (scores) at 12 weeks | baseline and up to 12 weeks
  Berg balance scale
change from baseline quality of life at 12 weeks | baseline and up to 12 weeks
  Pediatric Quality of Life inventory (PedsQL)

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Lan Hsieh, MD, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital; Taipei Medical University
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No